CLINICAL TRIAL: NCT03351543
Title: ADELE: Autoimmune Defense and Living Environment
Brief Title: Effect of Microbial Exposure on Health, Particularly Immune System
Acronym: ADELEWP1t4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Aki Sinkkonen, University researcher, docent, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HelsinkiUADELEWP1t4
Record Dates: First submitted 2016-03-23; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Immune System Disorders
Keywords: vaccine response; immune system activity
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposed group (Experimental): these volunteers receive microbial inoculate
  Interventions: Biological: microbial inoculate
- control (No Intervention): these volunteers do not receive microbial inoculate

INTERVENTIONS:
Biological: microbial inoculate — volunteers will regularly receive microbial inoculate that they do not use orally
  Arms: Exposed group

SUMMARY:
The effect of microbial exposure on healthy human subjects will be investigated. Changes in cytokine and IgE and vaccine response will be measured. The hypothesis is that microbial exposure increases the measured responses.

DETAILED DESCRIPTION:
The effect of microbial exposure on healthy human subjects will be investigated. The volunteers will either receive material containing a microbial inoculum, or they will receive nothing. Changes in cytokine and IgE and vaccine response will be measured. Subjective well-being will be recorded. Changes in microbial community will be followed. The hypothesis is that microbial exposure increases the measured responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults that live in urban conditions; that do not own a furry pet; that do not have HIV or other condition that weakens immune system; that do not use drugs chilling immune system; that do not have a history of five active infections that caused hospitalization within 2 years; that do not have a condition affecting immune response (e.g. rheumatoid, colitis ulcerosa, Crohn disease); that do not have dementia, acute depression or psychosis; that do not have cancer within 2 years; that do not have sore skin in arms or hands; that do not have diabetes; that do not have incompetency; that have not received earlier vaccine against Pneumococcus sp.; that do not have unwillingness to receive the vaccine; that do not live in countryside.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
difference in blood serum's cytokine levels | 1-3 months
  it will be checked if the values are different in different arms
difference in blood serum IgE levels | 1-3months
  in will be chekced if the values are different in different arms
Blood serum levels of antibodies caused by Prevenar 13 vaccine in different arms (intervention versus no intervention) | 1-3 months
  it will be checked if the values are different in different arms. Prevenar 13 is a vaccine against various Pneumococcus sp. infections

SECONDARY OUTCOMES:
difference in diversity (Shannon-Wiener index) of the composition of skin, stool and saliva bacterial community | 1-3 months
  it will be analyzed if microbial communities are similar in both arms
difference in richness (number of operational taxonomic units i.e. species) of the composition of skin, stool and saliva bacterial community | 1-3 months
  it will be analyzed if microbial communities are similar in both arms
Number of participants with treatment-related adverse events as assessed by a questionnaire described below | 1-3 months
  In the end of the experimental period and 2-4 weeks later, all study participants fill a questionnaire. It will be asked if the volunteers experienced a negative change in mental well-being during the study period. Similarly, they will be specifically asked for itches, skin symptoms and signs of infections. And index (how may yes-answers) will be compared between treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aki Sinkkonen, Ph D Docent, Study Chair — University of Helsinki
Locations (1):
- Helsinki University, Lahti, Kanta-Häme, Finland

IPD SHARING:
Plan to Share IPD: Yes
The data will be publicly available according to the instructions of Tekes, the funder. We can publish the data when we know the results and we have to publish it when the project ends.